CLINICAL TRIAL: NCT02502279
Title: Lung Recruitment and Postoperative CPAP in Pediatric Laparoscopic Surgery
Brief Title: Lung Recruitment and Postoperative CPAP
Acronym: LRvsCPAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, MD, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00008718/ refer.34
Record Dates: First submitted 2015-07-11; First posted 2015-07-20 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Engström Datex-Ohmeda ICU Ventilator: Pediatric patients under general anesthesia will be mechanically ventilated with the conventional ventilator parameters with 0 PEEP/CPAP.
- Lung Recruitment- PEEP group (Active Comparator): Engström Datex-Ohmeda ICU Ventilator: Pediatric patients under general anesthesia will be mechanically ventilated with the conventional ventilator parameters plus lung recruitment manoeuvre with peak inflation pressure 35 cmH2O for 15 seconds followed by PEEP until extubation delivered by the ventilator.
  Interventions: Device: Engström Datex-Ohmeda ICU Ventilator
- Lung Recruitment- PEEP and CPAP group (Active Comparator): Engström Datex-Ohmeda ICU Ventilator: Pediatric patients under general anesthesia will be mechanically ventilated with the conventional ventilator parameters plus
  1. lung recruitment manoeuvre with peak inflation pressure 35 cmH2O for 15 seconds followed by PEEP until extubation delivered by the ventilator.
  2. Postoperative CPAP mask immediately after extubation
  Interventions: Device: Engström Datex-Ohmeda ICU Ventilator; Device: Postoperative CPAP mask

INTERVENTIONS:
Device: Engström Datex-Ohmeda ICU Ventilator — patients will be mechanically ventilated and a vital capacity manoeuvre for lung inflation will be done by increasing the PIP to 35 cmH2o for 15 seconds followed by PEEP until extubation.
  Arms: Lung Recruitment- PEEP and CPAP group; Lung Recruitment- PEEP group
Device: Postoperative CPAP mask — patients will be mechanically ventilated and a vital capacity manoeuvre for lung inflation will be done by increasing the PIP to 35 cmH2o for 15 seconds followed by PEEP until extubation and a CPAP mask will be applied immediately postoperative.
  Arms: Lung Recruitment- PEEP and CPAP group

SUMMARY:
General anesthesia lowers FRC thereby promoting airway closure and absorption atelectasis. Alveolar recruitment manoeuvers recruit collapsed alveoli, increase gas exchange, and improve arterial oxygenation.

DETAILED DESCRIPTION:
General anesthesia lowers FRC thereby promoting airway closure and absorption atelectasis. Alveolar recruitment manoeuvers recruit collapsed alveoli, increase gas exchange, and improve arterial oxygenation. However, the effect of recruitment manoeuvre is short lasting and does not extend to the post operative period. Postoperative CPAP keeps the lung open and can improve oxygenation in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing laparoscopic surgery for abdominal cryptorchidism.

Exclusion Criteria:

* Cardio-respiratory illness.
* Unsatisfactory preoperative peripheral arterial oxygen saturation.
* Unsatisfactory preoperative hemoglobin level.
* Neurological or psychiatric disease.
* Children with a BMI >95th percentile for age.

Ages: 6 Months to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
(A-a) DO2 | 1 hour after extubation
  arterial blood gas will be withdrawn 1 hour after extubation and the alveolar minus arterial oxygen difference will be calculated for assessment of oxygenation

SECONDARY OUTCOMES:
PaO2 | intra-operative and 1hour postoperative
  arterial blood gas samples will be withdrawn to assess Pa O2.
PaCO2 | intra-operative and 1hour postoperative
  arterial blood gas samples will be withdrawn to assess PaCO2.
PH | intra-operative and 1hour postoperative
  arterial blood gas samples will be withdrawn to assess PH.
Respiratory mechanics | Intraoperative
  intra-operative ventilator data will be recorded to measure respiratory mechanics such as dynamic and statistic compliance
non invasive mean arterial pressure | intraoperative and 1hour postoperative
  non invasive mean arterial pressure will be recorded before and after recruitment manouvre, after pneumoperitonium and after pneumoperitonium deflation
Heart rate | intraoperative and 1hour postoperative
  the heart rate will be recorded before and after recruitment manoeuvre, after pneumoperitonium, and after pneumoperitonium deflation and early postoperative..
Peripheral arterial oxygenation SPO2% | intraoperative and 1hour postoperative
  The SPO2% will be recorded before and after recruitment manouvre, after peumoperitoneum inflation and after pneumoperitoneum deflation and early postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assisstant professor in Anesthesia and intensive care department, faculty of medicine, Assiut university, Egypt
Locations (1):
- Pediatric hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No